CLINICAL TRIAL: NCT04783558
Title: Effective Caregiving for Neonatal Abstinence Syndrome: Development of an Instructional Mobile Technology Platform for High-Risk Pregnant Women
Brief Title: Effective Caregiving for Neonatal Abstinence Syndrome: Testing an Instructional Mobile Technology Platform for High-Risk Pregnant Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Ekaterina Burduli, Assistant Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: K01DA051780 (NIH)
Record Dates: First submitted 2021-01-22; First posted 2021-03-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Neonatal Abstinence Syndrome; Opioid-use Disorder
MeSH Terms: conditions — Neonatal Abstinence Syndrome; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Pregnant women in the Treatment-as-Usual (TAU) condition will receive care as usual that involves continued enrollment in treatment and continued obstetric care. Participants will also be provided with a printed handout containing information on NAS and local resources. Pregnant women in the Adapted NAS tool Intervention will receive the adapted mobile-based NAS instructional tool and TAU. Women in this condition will go through the NAS instructional tool at least once during pregnancy, with their choice of going through the modules gradually while waiting at the OAT clinic to receive their dose, or by scheduling a time to review the modules. Participants will have free online access to the tool throughout their third trimester as well as through 12-weeks postpartum so they can access the modules at any time, and as many times as desired, including after giving birth. Women will be randomized 1:1 to the intervention or TAU conditions.
Masking Description: Women will be randomized 1:1 to the intervention or TAU conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted NAS tool Intervention (Experimental): Pregnant women in this condition will receive the adapted mobile-based NAS instructional tool and TAU. Women in this condition will go through the NAS instructional tool at least once during pregnancy, with their choice of going through the modules gradually while waiting at the OAT clinic to receive their dose, or by scheduling a time to review the modules. Participants will have free online access to the tool throughout their third trimester as well as through 12-weeks postpartum so they can access the modules at any time, and as many times as desired, including after giving birth.
  Interventions: Behavioral: Mobile-based NAS Caregiving Tool
- Treatment-as-Usual (TAU) (No Intervention): Pregnant women in this condition will receive care as usual that involves continued enrollment in OAT and continued obstetric care. We will also provide them with a printed handout containing information on NAS and local resources. Participants in the TAU condition will not receive iPads with accompanying modules, however the handout constitutes more information than they normally receive.

INTERVENTIONS:
Behavioral: Mobile-based NAS Caregiving Tool — The information and skills training in the adapted NAS caregiving tool will be largely based on elements of Eat Sleep Console. Therefore, the NAS mobile tool intervention will incorporate non-intrusive caregiving skills and strategies that encompass providing a low stimulating environment (e.g., dimmed light and low noise), swaddling, continuous comfort and contact with caregiver, skin-to-skin contact, frequent breastfeeding/feeding, as well as novel components identified in the key informant interviews (e.g., preparing for stigma during delivery, CPS involvement, etc.).
  Arms: Adapted NAS tool Intervention

SUMMARY:
Most newborns experiencing Neonatal Abstinence Syndrome (NAS) require non-pharmacologic care, which entails, most importantly, maternal involvement with her newborn. To facilitate positive maternal-newborn interactions, mothers need to learn effective caregiving NAS strategies while they are pregnant, yet, an enormous gap exists in the early education of mothers on the symptoms and progression of NAS, in part because no interventions exist to prepare future mothers for the challenges of caring for their newborns at risk for NAS. In this project, the investigators propose to adapt an existing mobile NAS tool for high-risk pregnant women and assess its usability, acceptability, and feasibility in a small randomized controlled analog trial.

DETAILED DESCRIPTION:
Due to an alarming rise in opioid use among the general population that is mirrored in pregnant women, Neonatal Abstinence Syndrome (NAS) rates have increased in the US from 2004 to 2014. Most newborns experiencing NAS require non-pharmacologic care, which entails, most importantly, maternal involvement with her newborn. Facilitating postpartum maternal-newborn involvement is critical in preventing further adverse maternal-newborn outcomes. To achieve positive maternal-newborn involvement, mothers need to learn effective caregiving NAS strategies while they are pregnant. Surprisingly, current obstetrical practice standards for high risk pregnant women do not address this pressing need, in part because no interventions exist to prepare future mothers for the challenges of caring for their newborns at risk for NAS. To address this critical gap, the investigators propose to adapt an existing mobile NAS tool for clinician training and decision support, for high-risk pregnant women and assess its usability, acceptability, and feasibility in a small randomized controlled analog trial. First, the investigators will conduct semi-structured interviews with a panel of neonatology experts, NAS care providers, and mothers with NAS-affected babies to gather their recommendations on management of NAS and explore their perspectives on the care of these newborns. Findings will guide the adaptation of the existing mobile NAS tool for high-risk pregnant women. The investigators will then test the usability, acceptability, and feasibility of the adapted mobile tool via surveys with 10 pregnant women receiving opioid agonist therapy (OAT) at Spokane Regional Health District's Opioid Treatment Program and Evergreen Recovery Center. Finally, the investigators will randomize 30 high-risk pregnant women seen at these facilities to either receive the adapted mobile NAS caregiving tool or usual care. The investigators will compare these mothers on maternal drug relapse and OAT continuation, maternal-newborn bonding, length of newborn hospital stays, readmission rates, breastfeeding initiation and duration, and postpartum depression and anxiety at 4, 8, and 12 weeks postpartum. Findings will serve as pilot data for a subsequent large R01 randomized controlled analog trial testing the efficacy of the adapted NAS caregiving tool in reducing poor outcomes for NAS-affected newborns and their mothers.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman in the third trimester currently in OAT treatment for opioid use disorder
* 18 years of age or older
* Ability to speak and understand English.

Exclusion Criteria:

• Recurring (e.g. daily or almost daily) thoughts of harming themselves or others in the past 2 weeks.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in maternal drug relapse | 4, 8, & 12 weeks postpartum
  Change will be assessed via the Addiction Severity Index-Lite (ASI-LITE), a standardized semi-structured clinical interview that offers clinical information and assesses severity profiles in the following domains: medical, employment, alcohol, drug, psychological, legal, and family/social.
Change in Opioid use treatment continuation | 4, 8, & 12 weeks postpartum
  Change in OAT continuation will be assessed via a direct question: "Are you currently receiving OAT (Y/N)? Please explain".

SECONDARY OUTCOMES:
Length of newborn hospital stay | 4, 8, & 12 weeks postpartum
  Length of newborn hospital stay will be assessed via a direct question: "how many days did your newborn stay in the hospital"
Newborn readmission | 4, 8, & 12 weeks postpartum
  Newborn hospital readmission will be assessed via direct questions at 3 time points: "has your newborn been readmitted to the hospital in the past 4 weeks for any reason? If yes, how many times in the past 4 weeks? Please list reasons for each readmission in the past 4 weeks"
maternal postpartum depression | 4, 8, & 12 weeks postpartum
  Maternal postpartum depression will be assessed via the PHQ-9, a psychometrically validated 9-item measure used to assess depression in a variety of populations. The PHQ-9 asks participants to report on the degree they were bothered by 9 symptoms over the past 2 weeks (i.e., "little interest or pleasure in doing things", "feeling down, depressed, or hopeless"), with response categories ranging from 0=not at all, to 3= nearly every day, and higher scores indicating greater levels of depression symptomology.
maternal postpartum stress | 4, 8, & 12 weeks postpartum
  Stress will be assessed via the Parenting Stress Index short form (PSI), which measures parental stress associated with the perception of having a difficult child or a dysfunctional parent-child relationship and consists of 36 items that are rated on a 5-point Likert scale (from 1-Strongly Agree to 5-Strongly Disagree) with higher scores indicative of less total stress. PSI has been shown to possess good psychometric properties and has been validated in numerous samples, including high-risk families. It includes Parental Distress, Parent-Child Dysfunctional Interaction and Difficult Child subscales, all of which will be considered individually. The Child and Parent domains can and will be combined to form a total stress scale score.
maternal-infant bonding | 4, 8, & 12 weeks postpartum
  Maternal-newborn bonding will be measured via the Maternal Postpartum Attachment Scale (MPAS.) It consists of 19 items assessing three dimensions: pleasure in interaction with the infant (5 items), absence of hostility towards the infant (5 items) and quality of mother-infant attachment (9 items). Response categories range from two-, three-, four- and five-point scales, for different items. The total score ranges from 19 to 95, with higher scores indicating higher maternal postpartum attachment to the baby. The MPAS has been found to have an acceptable level of reliability (Cronbach's alpha ranging from 0.75 to 0.79; test-retest reliability r= 0.86, p<.001).
breastfeeding | 4, 8, & 12 weeks postpartum
  Breastfeeding will be assessed via the following questions: "Are you currently breastfeeding? If yes, "How often do you breastfeed your baby?", if no, "How long did you breastfeed your baby"
maternal satisfaction with her birth experience | 4, 8, & 12 weeks postpartum
  To assess maternal satisfaction with her birth, the Birth Satisfaction Scale-Revised (BSS-R) will be used. The BSS-R is a 10-item, Likert-type, birth satisfaction questionnaire that measures experiences of childbearing, stress, quality of care, and women's attributes, and was psychometrically validated in the US. Its response categories range from 1 = Strongly Disagree, to 5 = Strongly Agree, with higher scores indicating higher birth satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington State University, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No
No individual level participant data will be shared with others.

REFERENCES:
- [Derived] Burduli E, Jones HE, Brooks O, Barbosa-Leiker C, Johnson RK, Roll J, McPherson SM. Development and Implementation of a Mobile Tool for High-Risk Pregnant Women to Deliver Effective Caregiving for Neonatal Abstinence Syndrome: Protocol for a Mixed Methods Study. JMIR Res Protoc. 2021 Apr 15;10(4):e27382. doi: 10.2196/27382. PMID 33856360